CLINICAL TRIAL: NCT06030258
Title: A Phase Ib/II Clinical Trial to Evaluate the Anti-tumor Efficacy, Safety, Tolerability, and Pharmacokinetics of IN10018 Combined With Anti-PD-1/L1 Antibody and Chemotherapy as First-line Treatment in Extensive-stage Small Cell Lung Cancer
Brief Title: IN10018 Combination Therapy in Treatment-naïve ES-SCLC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: InxMed (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN10018-019
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Small Cell Lung Cancer Extensive Stage
Keywords: First-line
MeSH Terms: interventions — tislelizumab; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): IN10018 in combination with Tislelizumab, carboplatin and etoposide as the first-line treatment in ES-SCLC.
  Interventions: Drug: IN10018; Drug: Tislelizumab; Drug: Carboplatin; Drug: Etoposide
- Control group (Active Comparator): Tislelizumab in combination with carboplatin and etoposide as the first-line treatment in ES-SCLC
  Interventions: Drug: Tislelizumab; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: IN10018 — orally taken once daily
  Other Names: BI 853520
  Arms: Experimental group
Drug: Tislelizumab — 200mg D1, Q3W, intravenously
Drug: Carboplatin — AUC 5 mg/ml/min, D1, Q3W, intravenously
Drug: Etoposide — Etoposide 100 mg/m2, D1-D3, Q3W, intravenously

SUMMARY:
This is a multicenter, open-label, Randomized, phase Ib/II clinical study to evaluate the anti-tumor efficacy, safety, tolerability, and PK of IN10018 in combination with anti-PD-1/L1 monoclonal antibody (Tislelizumab is proposed as the combination drug) and chemotherapy (platinum and etoposide) as the first-line treatment in Extensive-stage small cell lung cancer (ES-SCLC).

DETAILED DESCRIPTION:
This study consists of 2 parts: 1) Phase Ib-Dose Confirmation part: To assess the PK parameters, safety and recommended phase II dose (RP2D) of IN10018 in combination with anti-PD-1/L1 monoclonal antibody (Tislelizumab is proposed as the combination drug), platinum (carboplatin is proposed as the combination drug) and etoposide as the first-line treatment in ES-SCLC. 2) Phase II-Dose Expansion part: To assess the antitumor efficacy, safety and tolerability in the experimental group of IN10018 in combination with Tislelizumab, carboplatin and etoposide as compared to the control group of Tislelizumab in combination with carboplatin and etoposide as the first-line treatment in ES-SCLC.

ELIGIBILITY:
Inclusion Criteria

1. Male or female aged 18-75 years old at the time of signing informed consent.
2. Be able to understand and be willing to sign informed consent.
3. Histologically confirmed ES-SCLC (according to the Veterans Administration Lung Study Group (VALG) staging system), which is not suitable for locally radical therapy.
4. Has not received any systemic antitumor therapy for ES-SCLC.
5. Has at least one measurable tumor lesion per RECIST 1.1.
6. Has an ECOG performance status of 0 or 1.
7. Estimated life expectancy is more than 3 months.
8. Has adequate organ function of bone marrow, liver, kidney, and coagulation. Relative laboratory tests must be performed within 7 days prior to first dose of study treatment/randomization.
9. AEs due to prior antitumor therapy must be recovered to ≤ Grade 1 (CTCAE v5.0) or a steady state as assessed by investigators
10. Subjects (male and female) with childbearing potential must agree to use contraception during the treatment phase and through 3 months after the last dose of study treatment.

Exclusion Criteria

1. Has known active or untreated central nervous system (CNS) metastases, and/or carcinomatous meningitis.
2. Spinal cord compression without surgery and/or radiation therapy, or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for at least 7 days prior to the first dose of study treatment/randomization.
3. Pleural, pericardial or abdominal effusion that are clinically symptomatic and require puncture or drainage.
4. Symptomatic hypercalcemia.
5. Malignancies other than the study disease within 3 years prior to the first dose of study treatment/randomization.
6. Have received palliative radiotherapy for bone metastasis within 14 days prior to the first dose of study treatment/randomization.
7. Have had allogeneic haematopoietic stem cell transplantation or organ transplantation.
8. History of active autoimmune disease required systemic treatment (including but not limited to drugs for disease control, corticosteroids, or immunosuppressive drugs) within the past 2 years.
9. Have an immunodeficiency disorder or have received systemic steroid therapy (prednisone or equivalent corticosteroid > 10 mg/day) or other immunosuppressants within 7 days prior to the first dose of study treatment/randomization.
10. History of idiopathic pulmonary fibrosis, idiopathic pneumonia and organizing pneumonia, and interstitial pneumonitis or active pneumonia diagnosed per imaging examination at baseline.
11. Have had FAK inhibitors treatment.
12. Has a history of major cardiovascular or cerebrovascular diseases within 6 months prior to the first dose of study treatment/randomization.
13. Have malabsorption syndrome or cannot take study drugs orally.
14. Any active infection requiring systemic therapy within 14 days prior to the first dose of study treatment.
15. Active pulmonary tuberculosis
16. Human immunodeficiency virus (HIV) infection, active hepatitis B infection, or hepatitis C infection.
17. Known hypersensitivity or allergy to IN10018, anti-PD-1/L1 monoclonal antibodies, carboplatin or etoposide or to their drug components.
18. Pregnant or lactating women or are expected to be pregnant or lactating during study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-12-24 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
To identify the Recommended phase II dose (RP2D) of IN10018 in combination with Tislelizumab, Carboplatin and Etoposide in first-line ES-SCLC. | Up to 3 years
  Evaluate proportion of patients suffered with AEs defined as dose-limited toxicities (DLTs) per protocol; and RP2D will be determined per the incidence of AEs defined as DLTs.
Progress free survival (PFS) of IN10018 in combination with Tislelizumab, carboplatin and etoposide as compared to Tislelizumab in combination with carboplatin and etoposide in first-line ES-SCLC per BICR based on RECIST 1.1 | Up to 3 years
  Defined as the time from randomization to first documentation of disease progression or to death due to any cause, whichever comes first.

SECONDARY OUTCOMES:
PFS of IN10018 in combination with Tislelizumab, carboplatin and etoposide as compared to Tislelizumab in combination with carboplatin and etoposide in first-line ES-SCLC per investigator based on RECIST 1.1 | Up to 3 years
  Defined as the time from randomization to first documentation of disease progression or to death due to any cause, whichever comes first.
Objective response rate (ORR) of IN10018 in combination with Tislelizumab, carboplatin and etoposide as compared to Tislelizumab in combination with carboplatin and etoposide in first-line ES-SCLC per BICR and investigator based on RECIST 1.1. | Up to 3 years
  Defined as the proportion of subjects with complete response (CR) or partial response (PR).
Duration of objective response (DOR) of IN10018 in combination with Tislelizumab, carboplatin and etoposide as compared to Tislelizumab in combination with carboplatin and etoposide in first-line ES-SCLC per BICR and investigator based on RECIST 1.1. | Up to 3 years
  Defined as the time from start of the first documentation of CR or PR to the first documentation of disease progression or to death due to any cause, whichever comes first.
Disease Control Rate (DCR) of IN10018 in combination with Tislelizumab, carboplatin and etoposide as compared to Tislelizumab in combination with carboplatin and etoposide in first-line ES-SCLC per BICR and investigator based on RECIST 1.1 | Up to 3 years
  Defined as the proportion of patients with CR, PR, or stable disease (SD).
Overall survival (OS) of IN10018 in combination with Tislelizumab, carboplatin and etoposide as compared to Tislelizumab in combination with carboplatin and etoposide in first-line ES-SCLC. | Up to 3 years
  Defined as the time from randomization to the date of death due to any cause.
Number of patients with adverse event | Up to 3 years
  The number of participants who experienced AEs is presented.
PK: AUC of IN10018 following single dose administration and at steady state | Up to 3 years
  Area under the concentration-time curve (AUC)
PK: Cmax of IN10018 following single dose administration and at steady state | Up to 3 years
  Maximum concentration (Cmax)
PK: Ctrough of IN10018 following single dose administration and at steady state | Up to 3 years
  Trough concentration (Ctrough)
PK: Tmax of IN10018 following single dose administration and at steady state | Up to 3 years
  Time to Cmax (Tmax)
PK: t1/2 of IN10018 following single dose administration and at steady state | Up to 3 years
  Elimination half-life (t1/2)
PK: CL/F of IN10018 following single dose administration and at steady state | Up to 3 years
  apparent clearance (CL/F)
PK: Vd/F of IN10018 following single dose administration and at steady state | Up to 3 years
  Apparent volume of distribution (Vd/F)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhao, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (3):
- China (3):
  - Shandong Province Cancer Hospital, Jinan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Henan Provincial People's Hospital, Zhengzhou